CLINICAL TRIAL: NCT00962130
Title: Glucose Monitoring in Tissue Transfers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-2008-0066
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Reconstructive Tissue Surgery
Keywords: tissue perfusion; reconstructive surgery; continuous glucose monitoring
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood Glucose Measurement (Experimental): Subjects have sensors placed on skin before surgery and these sensors will measure the subject's glucose until the third day after surgery when they are removed.
  Interventions: Device: Continuous glucose monitoring system

INTERVENTIONS:
Device: Continuous glucose monitoring system — one or two monitors will be placed in the tissue to be transferred

SUMMARY:
The purpose of this study is to determine if 1) a continuous glucose monitoring system can measure glucose levels in transferred tissue during reconstructive surgery, and 2) if glucose measurements from a continuous glucose monitoring system correlate with tissue blood perfusion.

ELIGIBILITY:
Inclusion Criteria:

* presence of a soft tissue deformity where reconstruction with a pedicled or free tissue transfer is indicated
* age 18 and over
* ability to follow-up post-operatively

Exclusion Criteria:

* age less than 18
* prisoner status
* inability to participate in a standard post-operative follow-up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Perfusion and tissue transfer outcome during reconstructive surgery predicted by continuous glucose monitoring of tissue | Up to three days post-op

CONTACTS AND LOCATIONS:
Overall Officials: Timothy King, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States